CLINICAL TRIAL: NCT00720577
Title: Two-Part,Multicenter,Randomized,Double-Blind,Placebo-Controlled,Study to Evaluate the Effect of Simvastatin,Losartan,and Pioglitazone on Cardiovascular Disease Biomarkers in Lower Extremity Atherosclerotic Plaque Excised From Patients w/PAD
Brief Title: Study to Evaluate the Effect of Simvastatin, Losartan and Pioglitazone on Patients With Peripheral Arterial Disease.
Acronym: LEAP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Collaborators: FoxHollow Technologies (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FHT-P-05-005
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2008-07

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; PAD; Lower extremity peripheral arterial atherosclerotic plaque; RNA Expression; Lipid Biomarkers
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Simvastatin; Hydroxymethylglutaryl-CoA-Reductases, NADP-dependent; Losartan; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Simvastatin
- 2 (Active Comparator)
  Interventions: Drug: Losartan
- 3 (Active Comparator)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Simvastatin — 40 Mg. tablet, 1 tablet daily
  Other Names: HMG-CoA reductase
  Arms: 1
Drug: Losartan — 50 mg., tablets, 1 tablet once daily
  Other Names: Cozaar
  Arms: 2
Drug: Pioglitazone — 30 mg, tablet, 1 tablet once daily
  Other Names: Systematic (IUPAC)
  Arms: 3

SUMMARY:
Part A. The purpose of this study is to assess the effects of 6 weeks of treatment with, simvastatin, losartan or pioglitazone compared to placebo on the RNA expression profile of lower extremity peripheral arterial atherosclerotic plaque. Part B. The effect of simvastatin, losartan or pioglitazone compared to placebo on protein and lipid biomarkers in lower extremity peripheral arterial atherosclerotic plaque.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, 6 week study. The study consists of 3 separate sub-studies in which patients undergoing bilateral lower extremity peripheral artery atherectomy will receive one of three FDA approved drugs known to have beneficial effect on the risk of cardiovascular disease. Patients will be selected for the particular sub-study based on a series of entry criteria and then randomized to the particular agent or placebo for 6-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women =90 years of age.
* Bilateral lower extremity PAD requiring revascularization. Both extremities must have at least 1denovo atherosclerotic lesion
* Able to space bilateral atherectomy procedures by at least 6 weeks.
* Willing to provide informed consent to participation in genetic studies.
* Simvastatin Substudy
* LDL-C >100 mg/dL and <250 mg/dL TG<350 mg/dL
* Not currently receiving or having taken a statin (simvastatin, lovastatin, rosuvastatin, atorvastatin, or pravastatin) or a combination product containing a statin for the previous 3 months.
* Losartan Substudy
* Diagnosis of hypertension with systolic blood pressure >120 mm Hg but <160 mm Hg, and diastolic blood pressure >80 mm Hg but <100 mm Hg.
* Not currently receiving or having taken an ACEi or ARB.
* Pioglitazone Substudy
* Type II diabetes mellitus
* HbA1c >5.5% and < 8.5%
* Otherwise on a stable glucose lowering regimen where no changes are expected in oral regimen, or where no changes in insulin doses of more than 10 U are expected.
* Not currently receiving or having taken a thiazolidinedione (rosiglitazone or pioglitazone) or a combination product containing a thiazolidinedione or the previous 12 months.

Exclusion Criteria:

* Patient is pregnant, breast-feeding, or expecting to conceive during the study including the 14-day post study follow-up.
* current condition, therapy, lab abnormality, mental legal incapacitation that in the investigator's judgment might confound the results of the study.
* Patient is currently participating in or has participated in a study with an investigational compound within 30 days of Visit 1.
* Patient has donated and/or received blood (including phlebotomy of >300 mL) within 2 months prior to study.
* Surgery or significant trauma within 2 months prior to Visit 1.
* Patient is a user of recreational or illicit drugs or has had a recent history <1yr drug/alcohol abuse>2 alcoholic drinks per day).
* Patient was <80% compliant with dosing during the placebo run-in period AND, in the opinion of the investigator, believed to be unable to maintain at least an 80% compliance with dosing during the active study dosing period.
* Patient has history of myocardial infarction, stroke, coronary artery bypass surgery or other coronary, carotid, or cerebral revascularization procedure,unstable angina, or angioplasty within 1 month of Visit 1. - Patient has chronic heart failure defined by New York Heart Association NYHA) Classes III or IV.
* Known clinically significant AV conduction disturbances or arrhythmias
* Patient has unstable hypertension (e.g., sitting systolic blood pressure >160 mm Hg or diastolic >100 mm Hg) at Visit 1.
* Any known clinically important bleeding or platelet disorder.
* Patient has history of ileal bypass, gastric bypass, other significant condition associated with malabsorption.
* Patient is HIV or hepatitis B positive.
* Patients with significantly elevated TSH at Visit 1 may be entered after consultation with and approval by the SPONSOR. Patients with a history of hypothyroidism, who are on a stable dose of thyroxine with normal TSH level at Visit 1 may be included.
* Patients on cyclical estrogen medications (Estrogen Replacement Therapy ERT] or oral contraceptives). Patients on non-cyclical estrogen replacement therapy or Selective Estrogen Receptor Modulator (SERM) may be included, but must be on a stable dose for at least 8 weeks prior.
* Patients with active neoplastic disease which compromises their general health, or who currently require chemotherapy or radiation therapy, or who have completed chemotherapy or radiation therapy within 3 months prior.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Evaluate RNA expression profiles, protein and lipid biomarkers, and gene expression profiling on pts receiving simvastatin, losartan or pioglitazone. | 6 weeks

SECONDARY OUTCOMES:
Evaluate plaque characteristics in 3 patient subsets and Left and Right extremity comparisons. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Duke University